CLINICAL TRIAL: NCT05798624
Title: To Study the Impact of a Previous Cesarean Section (CS) With / Without an Isthmocele on the Ongoing Pregnancy Rate in Single Euploid Frozen Embryo Transfer
Brief Title: Impact of a Previous CS on the Ongoing Pregnancy Rate in Single Euploid Frozen Embryo Transfer (ET)
Status: Recruiting | Type: Observational
Sponsor: ART Fertility Clinics LLC (Other)
Responsible Party: Principal Investigator, Barbara Lawrenz, Scientific Director, ART Fertility Clinics LLC
Other Study IDs: 2303-ABU-003-BL
Record Dates: First submitted 2023-03-23; First posted 2023-04-04 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-07

CONDITIONS: Infertility; Implantation
Keywords: Implantation; Infertility; Isthmocele; Cesarean section
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- One CS with isthmocele
  Interventions: Diagnostic Test: Ultrasound between 6+0 and 6+7 weeks of pregnancy - With Isthmocele
- More than one CS with Isthmocele
  Interventions: Diagnostic Test: Ultrasound between 6+0 and 6+7 weeks of pregnancy - With Isthmocele
- One or more CS without isthmocele
  Interventions: Diagnostic Test: Ultrasound between 6+0 and 6+7 weeks of pregnancy - Without Isthmocele
- With previous vaginal delivery
  Interventions: Diagnostic Test: Ultrasound between 6+0 and 6+7 weeks of pregnancy
- With first ongoing pregnancy
  Interventions: Diagnostic Test: Ultrasound between 6+0 and 6+7 weeks of pregnancy

INTERVENTIONS:
Diagnostic Test: Ultrasound between 6+0 and 6+7 weeks of pregnancy - With Isthmocele — Location of implantation of the GS (gestational sac) amended to Naji et al, defined as 3 possible implantation sites: (A: fundal, B: anterior, C: posterior)
  Size of isthmocele:
  * Depth of isthmocele
  * Width of isthmocele
  * Circumference of isthmocele
  Distance between isthmocele and outer cervical os (measured with the trace line) Distance between CS scar and outer cervical os (measured with the trace line) Size of gestational sac Measurements of the isthmocele size / circumference / distance between isthmocele / CS and outer cervical os
  Groups: More than one CS with Isthmocele; One CS with isthmocele
Diagnostic Test: Ultrasound between 6+0 and 6+7 weeks of pregnancy - Without Isthmocele — Location of implantation of the GS amended to Naji et al, defined as 3 possible implantation sites: (A: fundal, B: anterior, C: posterior) Distance between CS scar and outer cervical os (measured with the trace line) Size of gestational sac
  Groups: One or more CS without isthmocele
Diagnostic Test: Ultrasound between 6+0 and 6+7 weeks of pregnancy — Location of implantation of the GS (gestational sac) amended to Naji et al, defined as 3 possible implantation sites (A: fundal, B: anterior, C: posterior)
  Size of gestational sac
  Groups: With first ongoing pregnancy; With previous vaginal delivery

SUMMARY:
As embryo ploidy is a crucial factor not only for implantation but also for maintenance of a pregnancy, the aim of this study is to evaluate the impact of the CS / isthmocele on the ongoing pregnancy rates and the implantation site in single euploid frozen embryo transfer, independent of the endometrial preparation approach.

DETAILED DESCRIPTION:
The impact of a previous CS on the future fertility in the general population is discussed controversially, but it seems that the clinical and social circumstances leading to the CS have a greater effect on future fertility than the surgical procedure itself (Gurol-Urganci et al., 2013, 2014; Evers et al., 2014). However, this might be different in women who do not conceive spontaneously after a previous CS and need to undergo ART due to secondary infertility. Whereas some studies describe a reduction of implantation, ongoing pregnancy, and live birth (LB) rates (Vissers et al., 2020; Wang et al., 2020; Diao et al., 2021; Friedenthal et al., 2021; van den Tweel et al., 2022), others describe a negative impact of a previous CS only in the presence of an isthmocele (Diao et al., 2021) or no impact (Patounakis et al., 2016).

A case control study evaluated whether there are any differences in the location and distance to the internal cervical ostium of the implantation site of the intrauterine gestation sacs, early pregnancy symptoms and pregnancy outcome at 12 weeks gestation between women with and without a previous Caesarean section (CS) in patients who conceived naturally (Naji et al., 2013). Investigators concluded that the presence of a CS scar affects the site of implantation, and also that the distance between implantation site and the scar is related to the risk of spontaneous abortion.

This is a purely observational study without any intervention. Participants will be stratified into different groups according to their previous obstetrical history. Total sample size will include 1050 participants undergoing a frozen embryo transfer (FET) cycle.

Isthmocele will be defined according to de Vaate et al (Bij de Vaate et al., 2011) as: visible anechogenic area of at least 1 mm depth at the site of the Cesarean scar.

ELIGIBILITY:
Inclusion Criteria:

- All participants undergoing a single euploid FET, independent of the endometrial preparation approach

Exclusion Criteria:

* Intracavitary fluid during preparation for FET
* Known anomaly of the uterus or the adnexae (e.g.: fibroids, polyps, hydrosalpinx, endometriosis, adenomyosis)
* Embryo which was biopsied on day 7
* Poor quality embryo which was transferred (Gardner criteria: AC / BC / CB, biopsied on day 6 and CC embryos from both, day 5 and day 6 biopsies, classified as "poor" quality embryos)
* History of recurrent abortion
* Antiphospholipid syndrome / autoimmune diseases

Ages: 18 Years to 42 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes
Study Population: Female undergoing IVF/ICSI treatment
Sampling Method: Non-Probability Sample
Enrollment: 1050 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2025-05-15 (Estimated); Study Completion 2025-07-30 (Estimated)

PRIMARY OUTCOMES:
Ongoing pregnancy rate | 5 weeks
Implantation rate | 6 weeks
  Number of gestational sacs observed by ultrasound at 6 weeks of gestation divided by the number of embryos transferred
Implantation site | 6 weeks
Rate of vaginal bleeding in early pregnancy (until 12 weeks of gestation) | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Lawrenz, PhD, Principal Investigator — ART Fertility Clinics LLC
Locations (1):
- ART Fertility Clinics LLC, Abu Dhabi, United Arab Emirates

REFERENCES:
- [Background] Betran AP, Ye J, Moller AB, Souza JP, Zhang J. Trends and projections of caesarean section rates: global and regional estimates. BMJ Glob Health. 2021 Jun;6(6):e005671. doi: 10.1136/bmjgh-2021-005671. PMID 34130991
- [Background] Bij de Vaate AJ, Brolmann HA, van der Voet LF, van der Slikke JW, Veersema S, Huirne JA. Ultrasound evaluation of the Cesarean scar: relation between a niche and postmenstrual spotting. Ultrasound Obstet Gynecol. 2011 Jan;37(1):93-9. doi: 10.1002/uog.8864. PMID 21031351
- [Background] Diao J, Gao G, Zhang Y, Wang X, Zhang Y, Han Y, Du A, Luo H. Caesarean section defects may affect pregnancy outcomes after in vitro fertilization-embryo transfer: a retrospective study. BMC Pregnancy Childbirth. 2021 Jul 6;21(1):487. doi: 10.1186/s12884-021-03955-7. PMID 34229640
- [Background] Evers EC, McDermott KC, Blomquist JL, Handa VL. Mode of delivery and subsequent fertility. Hum Reprod. 2014 Nov;29(11):2569-74. doi: 10.1093/humrep/deu197. Epub 2014 Aug 27. PMID 25164023
- [Background] Friedenthal J, Alkon-Meadows T, Hernandez-Nieto C, Gounko D, Lee JA, Copperman A, Buyuk E. The association between prior cesarean delivery and subsequent in vitro fertilization outcomes in women undergoing autologous, frozen-thawed single euploid embryo transfer. Am J Obstet Gynecol. 2021 Sep;225(3):287.e1-287.e8. doi: 10.1016/j.ajog.2021.03.026. Epub 2021 Mar 30. PMID 33798478
- [Background] Gurol-Urganci I, Bou-Antoun S, Lim CP, Cromwell DA, Mahmood TA, Templeton A, van der Meulen JH. Impact of Caesarean section on subsequent fertility: a systematic review and meta-analysis. Hum Reprod. 2013 Jul;28(7):1943-52. doi: 10.1093/humrep/det130. Epub 2013 May 3. PMID 23644593
- [Background] Gurol-Urganci I, Cromwell DA, Mahmood TA, van der Meulen JH, Templeton A. A population-based cohort study of the effect of Caesarean section on subsequent fertility. Hum Reprod. 2014 Jun;29(6):1320-6. doi: 10.1093/humrep/deu057. Epub 2014 Apr 29. PMID 24781430
- [Background] Lawrenz B, Melado L, Garrido N, Coughlan C, Markova D, Fatemi H. Isthmocele and ovarian stimulation for IVF: considerations for a reproductive medicine specialist. Hum Reprod. 2020 Jan 1;35(1):89-99. doi: 10.1093/humrep/dez241. PMID 31885047
- [Background] Naji O, Wynants L, Smith A, Abdallah Y, Saso S, Stalder C, Van Huffel S, Ghaem-Maghami S, Van Calster B, Timmerman D, Bourne T. Does the presence of a Caesarean section scar affect implantation site and early pregnancy outcome in women attending an early pregnancy assessment unit? Hum Reprod. 2013 Jun;28(6):1489-96. doi: 10.1093/humrep/det110. Epub 2013 Apr 12. PMID 23585560
- [Background] Patounakis G, Ozcan MC, Chason RJ, Norian JM, Payson M, DeCherney AH, Yauger BJ. Impact of a prior cesarean delivery on embryo transfer: a prospective study. Fertil Steril. 2016 Aug;106(2):311-6. doi: 10.1016/j.fertnstert.2016.03.045. Epub 2016 Apr 14. PMID 27087400
- [Background] Sandall J, Tribe RM, Avery L, Mola G, Visser GH, Homer CS, Gibbons D, Kelly NM, Kennedy HP, Kidanto H, Taylor P, Temmerman M. Short-term and long-term effects of caesarean section on the health of women and children. Lancet. 2018 Oct 13;392(10155):1349-1357. doi: 10.1016/S0140-6736(18)31930-5. PMID 30322585
- [Background] van den Tweel MM, Klijn NF, Diaz de Pool JDN, van der Westerlaken LAJ, Louwe LA. Previous caesarean section is associated with lower subsequent in vitro fertilization live birth rates. Hum Fertil (Camb). 2022 Feb;25(1):93-98. doi: 10.1080/14647273.2019.1696990. Epub 2019 Dec 3. PMID 31793367
- [Background] Vissers J, Sluckin TC, van Driel-Delprat CCR, Schats R, Groot CJM, Lambalk CB, Twisk JWR, Huirne JAF. Reduced pregnancy and live birth rates after in vitro fertilization in women with previous Caesarean section: a retrospective cohort study. Hum Reprod. 2020 Mar 27;35(3):595-604. doi: 10.1093/humrep/dez295. PMID 32142117
- [Background] Wang L, Yao W, Tang X, Yao H, Wei S, Huang J, Mol BWJ, Jin L, Yue J, Wang R. Fertility outcomes of IVF/ICSI after Caesarean section: a cohort study. Reprod Biomed Online. 2020 May;40(5):719-728. doi: 10.1016/j.rbmo.2019.12.004. Epub 2019 Dec 16. PMID 32336649